CLINICAL TRIAL: NCT01536795
Title: Topical Treatment of Old World Cutaneous Leishmaniasis With WR279396 (Paromomycin/Gentamicin Ointment): Efficacy and Tolerance of a Regimen Using an Occlusive Polyurethane Dressing
Brief Title: A Study to Evaluate the Efficacy and Tolerance of WR279,396 for Old World Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-9768.2; IND50,098 (Other: US FDA)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2021-01-07 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Old World Cutaneous Leishmaniasis
Keywords: Ointment to treat leishmania skin lesions
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- WR279,396 with Tegaderm dressing (Experimental): 24 patients will be randomly allocated to WR279,396 treatment once-a-day for 20 days with using an occlusive polyurethane Tegaderm dressing
  Interventions: Drug: WR279,396 with Tegaderm Dressing
- WR279,396 with Gauze and Tape Dressing (Experimental): 24 subjects will be randomly allocated to WR279,396 treatment once a day for 20 days without an optimized polyurethane dressing (gauze and tape only).
  Interventions: Drug: WR 279,396 with Gauze and Tape Dressing

INTERVENTIONS:
Drug: WR279,396 with Tegaderm Dressing — Ointment containing paromomycin sulphate (15%) and gentamicin sulphate (0.5%) - in a base (AQIC)applied for 20 days with polyurethane dressing
  Arms: WR279,396 with Tegaderm dressing
Drug: WR 279,396 with Gauze and Tape Dressing — Ointment containing paromomycin sulphate (15%) and gentamicin sulphate (0.5%) - in a base (AQIC)applied for 20 days
  Arms: WR279,396 with Gauze and Tape Dressing

SUMMARY:
This Phase 2 study is to determine whether WR279396 with occlusion (a polyurethane dressing) is more effective than WR279396 without occlusion for once daily treatment.

Extensive objective and subjective local tolerance data will also be captured during this trial, as well as surrogate markers (parasite loads and aminoglycosides concentration in the deep dermis) that may help to determine the optimal number and duration of treatments.

The results from this study will help determine the most practical treatment schedule and will answer questions that are crucial to improve the present treatment regimen with WR279396 which is twice a day for 20 days.

DETAILED DESCRIPTION:
Forty-eight patients (48) with Old World cutaneous leishmaniasis will be randomly allocated to WR279396 treatment once a day for 20 days with an optimized polyurethane dressing (occlusion) (24 patients), or without occlusion (24 patients). All patients will be rescued with the standard of care accepted in Tunisia, if the patient is not cured. The active ingredients of WR279396 are two aminoglycosides - paromomycin sulphate (15%) and gentamicin sulphate (0.5%) - in a base (AQIC).

Each subject will be followed for clinical cure for 90 days after the initiation of treatment. Cure is defined as 100% reepithelialization without relapse by 3 months.

Tolerance will be evaluated by local adverse reactions and by laboratory signs of systemic events.

In addition to the clinical evaluation of the CL lesions, the following parameters/clinical healing surrogates will be investigated:

1. parasite load will be determined in superficial and deep lesional dermis samples at D0 and D10. The mean parasite reduction ratio (parasite load at D10/parasite load at D0) in each group will be compared;
2. aminoglycoside concentrations in superficial and deep infiltrated dermis in each group will be compared.

ELIGIBILITY:
Inclusion Criteria: The study population will be selected from adults (18y) patients and children above 15y in Tunisia (Old World)

* Age: 15 - 75 years old
* Lesion character: each diameter (horizontal and vertical) of the lesion test must measure 7 mm, the lesion must be primarily ulcerative (i.e., not verrucous or nodular) and located in a biopsy friendly site of the body
* Parasitological diagnosis: have cutaneous leishmaniasis proven parasitologically in lesion selected for inclusion in study (lesion test).
* Informed consent: have given written informed consent to participate in the study: (i.e. patient or legal representative).

Exclusion Criteria:

* Drug intolerance: history of known or suspected hypersensitivity or idiosyncratic reactions to aminoglycosides in the patient or immediate family members.
* Previous use of antileishmanial drugs (within 2 months) or present use of routinely nephrotoxic or ototoxic drugs.
* Potential for follow up: Have less than 4 months time remaining in present address and/or plans to leave the area for more than 30 days.
* Extent of disease: More than 10 lesions or lesion ³ 5 cm or a lesion less than 2 cm from eye, in the ear, or a lesion in the face, that in the opinion of the attending dermatologist could potentially cause significant disfigurement.
* Location of disease: mucosal involvement.
* Disseminated disease: clinically significant lymphadenitis with nodules that are painful and > 1 cm in size in the lymphatic drainage of the ulcer.
* Concomitant medical problems: significant medical problems of the kidney or liver as determined by history and by the following laboratory studies:
* Kidney: clinically significant abnormalities of urine analysis, serum levels of Creatinine, BUN, total proteins > upper limit of normal for the laboratory.
* Liver: AST or ALT > upper limit of normal for the laboratory.
* General: glucose, Na, K, > upper limit of normal or < lower limit of normal for the laboratory. Volunteers in whom these normal laboratory values are exceeded by less than 25% will not be automatically excluded. These volunteers will be evaluated on the basis of history, physical, as well as laboratory values.
* Scheduled or ongoing pregnancy as determined clinical and biological criteria.
* Presence of signs or symptoms of peripheral neuropathy, myasthenia gravis or neuromuscular block

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afif Ben Salah,, MD, PhD, Principal Investigator — Institut Pasteur, Tunisia
Locations (1):
- Institut Pasteur, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 48 subjects were randomized and received treatment at the Institut Pasteur de Tunis and primary healthcare centers and schools of the study area in Sidi Bouzid and Elmmara, Tunisia.
Period: Overall Study
Arm/Group | WR279,396 With Tegaderm Dressing | WR279,396 With Gauze and Tape Dressing
Started | 24 | 24
Completed | 23 | 22
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WR279,396 With Tegaderm Dressing | WR279,396 With Gauze and Tape Dressing | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 5 | 11
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 12 | 11 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Middle Eastern or North African | 24 | 23 | 47
  Race: Other (European/Arab) | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Tunisia | 24 | 24 | 48
Subjects with a previous history of leishmaniasis [Count of Participants; unit: Participants]
  Yes | 3 | 2 | 5
  No | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Safety: Overview of Adverse Events
Description: Safety of WR279,396 through the tracking of local, systemic and spontaneous adverse reactions
Time Frame: During 20 day treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | WR279,396 With Tegaderm Dressing | WR279,396 With Gauze and Tape Dressing
Number analyzed (Participants) | 24 | 24
Participants
  Subjects with atleast 1 AE | 16 | 7
  Subjects with an SAE | 0 | 0
  Withdrawals due to an AE | 0 | 0
  Not due to an AE | 0 | 1
  Deaths | 0 | 0

2. Secondary Outcome: Clinical Responses of Index Lesions (100% Re-epithelialization)
Description: Efficacy will be evaluated in terms of the number of lesions cured at D50 (D1 is the first day of treatment) with no relapse by Day 90. Complete clinical respoonse is defined as 100% re-epithelialization of the index lesion by Day 50 or a > 50% re-epithelialization by Day 50 followed by complete re-epithelialization on or before Day 90, with no relapse ever having occurred from Day 50 through Day 90.
Time Frame: Day 50, 90
Measure: Count of Participants; unit: Participants
Arm/Group | WR279,396 With Tegaderm Dressing | WR279,396 With Gauze and Tape Dressing
Number analyzed (Participants) | 24 | 24
Participants
  Day 50 - Not Evaluable | 1 | 2
  Day 50 - Cured | 19 | 20
  Day 50 - Improved | 2 | 2
  Day 50 - Failure | 2 | 0
  Day 90 - Not Evaluable | 1 | 2
  Day 90 - Cured/Improved at D50 with no relapse | 17 | 20
  Day 90 - Improved | 2 | 2
  Day 90 - Failure | 4 | 0

3. Other Pre Specified Outcome: Area of the Index Lesion's Ulceration by Study Day
Description: Area of the index lesion's ulceration over time in mm2
Time Frame: Days 1, 10, 20, 50 and 90
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | WR279,396 With Tegaderm Dressing | WR279,396 With Gauze and Tape Dressing
Number analyzed (Participants) | 24 | 24
mm^2
  Day 0/1 | 127.0 (147.39) | 157.69 (179.52)
  Day 10 | 118.87 (106.41) | 140.64 (157.74)
  Day 20 | 115.62 (101.45) | 153.51 (176.37)
  Day 50 | 20.0 (48.3) | 1.3 (6.2)
  Day 90 | 30.8 (117.9) | 0.00 (0.0)

4. Other Pre Specified Outcome: Area of the Index Lesion's Induration by Study Day
Description: Area of the index lesion's induration over time in mm2
Time Frame: Days 1, 10, 20, 50 and 90
Population: On D50 in the Gauze-Tape group no SD was given in the data table. All good cause efforts to locate the data for Day 50 SD value for gauze and tape dressing arm have been exhausted, data are missing and hence not available to be reported.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | WR279,396 With Tegaderm Dressing | WR279,396 With Gauze and Tape Dressing
Number analyzed (Participants) | 24 | 24
mm^2
  Day 0/1 | 360.7 (262.5) | 505.9 (431.6)
  Day 10 | 405.14 (250.78) | 495.25 (401.47)
  Day 20 | 410.15 (269.62) | 468.85 (344.01)
  Day 50 | 122.7 (249.8) | 148.05 (NA) — All good cause efforts to locate the data have been exhausted, data are missing and hence not available to be reported.
  Day 90 | 74.6 (235.4) | 0.00 (0.00)

5. Other Pre Specified Outcome: Percentage Change in Induration Area From Baseline and Days 10, 20, 50 and 90
Description: Percentage of change of index lesion in induration area from baseline and days 10, 20, 50 and 90
Time Frame: Days 10, 20, 50 and 90
Measure: Mean (Standard Deviation); unit: % change in induration
Arm/Group | WR279,396 With Tegaderm Dressing | WR279,396 With Gauze and Tape Dressing
Number analyzed (Participants) | 24 | 24
% change in induration
  Day 10 | 28.3 (63.2) | 45.0 (114.2)
  Day 20 | 30.0 (62.0) | 51.0 (116.2)
  Day 50 | -64.4 (78.5) | -83.9 (30.7)
  Day 90 | -65.1 (98.5) | -100.0 (0)

ADVERSE EVENTS:
Time Frame: 90 Days
Arm/Group | WR279,396 With Tegaderm Dressing | WR279,396 With Gauze and Tape Dressing
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 16/24 | 7/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WR279,396 With Tegaderm Dressing (N=24) | WR279,396 With Gauze and Tape Dressing (N=24)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Local reaction (infection at biopsy site) (General disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 1 (1) | 5 (5)
Pain (General disorders) | 1 (1) | 4 (4)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Any infection and infestation (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Any investigations (Investigations) | 4 (4) | 1 (1)
Blood creatinine increased (Investigations) | 4 (4) | 1 (1)
Blister (vesicles) (Skin and subcutaneous tissue disorders) | 10 (10) | 3 (3)
Dermatitis contact (allergy to Tegaderm) (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No